CLINICAL TRIAL: NCT07050329
Title: Comparison of Outcome With Ultrasonic Dissector Versus Electrocautery in Modified Radical Mastectomy
Brief Title: Comparison of Operation Time, Drain Duration, and Seroma Formation After Modified Radical Mastectomy Using Ultrasonic Dissector Versus Electrocautery in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quaid-e-Azam Medical College (Other)
Responsible Party: Principal Investigator, Dr.Maryum Naveed, Principal Investigator, Quaid-e-Azam Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1324-5017
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Mastectomy, Modified Radical; Mastectomy Plus Axillary Lymph Node Dissection; Seroma Following Procedure
Keywords: Breast carcinoma; electrocautery; modified radical mastectomy; ultrasonic dissector; axillary dissection; post-mastectomy seroma; Bipolar electrocautery
MeSH Terms: conditions — Breast Neoplasms | interventions — Electrocoagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrocautery Dissection Group (Active Comparator): Axillary dissection was performed as per standard hospital protocol.
  Interventions: Device: Electrocautery
- Ultrasonic Dissection Group (Experimental): Axillary dissection was performed using ultrasonic dissector.
  Interventions: Device: Ultrasonic dissector

INTERVENTIONS:
Device: Electrocautery — Axillary dissection was done through bipolar electrocautery
  Other Names: Bipolar electrocautery
  Arms: Electrocautery Dissection Group
Device: Ultrasonic dissector — Axillary dissection was done through ultrasonic dissector.
  Arms: Ultrasonic Dissection Group

SUMMARY:
The goal of this clinical trial was to compare two surgical techniques-ultrasonic dissector and electrocautery-for performing axillary dissection in women undergoing modified radical mastectomy (MRM) for breast cancer. The study aimed to determine whether using an ultrasonic dissector reduces operation time, the number of days surgical drains remain in place, and the frequency of seroma formation compared to conventional electrocautery.

The main questions the study aims to answer are:

1. Does the ultrasonic dissector reduce the duration of surgery compared to electrocautery?
2. Do patients operated with an ultrasonic dissector require surgical drains for fewer days?
3. Is the frequency of postoperative seroma formation lower in the ultrasonic dissector group?

Researchers randomly (1:1) assigned 138 women with breast cancer (aged 35-65 years) undergoing MRM to either the ultrasonic dissector group or the electrocautery group. All surgeries were performed by experienced consultant surgeons using standardized protocols.

Participants:

* Underwent MRM with either electrocautery or ultrasonic dissector for axillary dissection
* Were discharged 24 hours after surgery with two drains in place
* Measured and reported daily drain output at home
* Returned for weekly follow-up for 30 days postoperatively

Outcomes were measured by recording the operation time, the number of days drains remained in place, and the occurrence of seroma. The results would help guide surgical practice by identifying the safer and more efficient dissection method during MRM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer and
* Planned for modified radical mastectomy

Exclusion Criteria:

* Planned with immediate reconstruction
* Women with recurrent breast cancer and
* Women with previous radiation over chest wall

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Seroma Formation | 30 days postoperatively
  Presence of fluid collection beneath the skin flaps after the removal of the drains of sufficient quantity to cause the patient discomfort and was measured by subcutaneous aspiration & through ultrasonography during the postoperative follow up

OTHER OUTCOMES:
Surgery Time | Intraoperative
  Duration (minutes) of surgery was noted from skin incision to skin closure using stopwatch.
Drains Duration | 30 days postoperatively
  Time in days from placement to removal of drain will be calculated. The drains will be removed when the drainage volume is less than 30 ml over 24 h for 2 successive days.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq I Professor, FCPS, Study Chair — Quaid-e-Azam Medical College
Locations (1):
- Quaid-e-Azam Medical College, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayer JH. Slide reproduction of radiographs: improved results with color film. AJR Am J Roentgenol. 1982 Feb;138(2):361-2. doi: 10.2214/ajr.138.2.361. No abstract available. PMID 6976748
- [Background] Deori A, Gupta N, Gupta AK, Yelamanchi R, Agrawal H, Durga CK. A Prospective Randomised Controlled Study Comparing Ultrasonic Dissector with Electrocautery for Axillary Dissection in Patients of Carcinoma Breast. Malays J Med Sci. 2021 Feb;28(1):97-104. doi: 10.21315/mjms2021.28.1.12. Epub 2021 Feb 24. PMID 33679225